CLINICAL TRIAL: NCT00818441
Title: A PHASE 2, OPEN-LABEL TRIAL OF DACOMITINIB (PF-00299804) IN SELECTED PATIENTS WITH ADVANCED ADENOCARCINOMA OF THE LUNG
Brief Title: Dacomitinib (PF-00299804) As A Single Oral Agent In Selected Patients With Adenocarcinoma Of The Lung
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: A7471017; 2011-002794-39 (EudraCT Number)
Record Dates: First submitted 2009-01-05; First posted 2009-01-07 (Estimated); Results first posted 2016-06-01 (Estimated); Last update posted 2019-01-08 (Actual); Status verified 2018-12

CONDITIONS: Carcinoma, Non-small Cell
Keywords: lung cancer adenocarcinoma HER2
MeSH Terms: conditions — Carcinoma | interventions — dacomitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort A (Experimental): Dacomitinib (PF-00299804) in patients with EGFR mutated NSCLC or clinical characteristics defined above to enhance for EGFR mutated NSCLC
  Interventions: Drug: Dacomitinib (PF-00299804)
- Cohort B (Experimental): Dacomitinib in patients with HER2 mutated or amplified NSCLC
  Interventions: Drug: Dacomitinib (PF-00299804)

INTERVENTIONS:
Drug: Dacomitinib (PF-00299804) — Dacomitinib (PF-00299804) at 45 mg daily or 30 mg daily by continuous oral dosing, to be escalated in tolerating patients to 45mg after at least 8 weeks of therapy (30 patients in Cohort A started at the lower dose).
  Arms: Cohort A
Drug: Dacomitinib (PF-00299804) — In Cohort B, patients getting Dacomitinib for first line therapy started at 30 mg, but those who had prior anti-cancer therapy started at 45 mg.
  Arms: Cohort B

SUMMARY:
This study will explore the safety and efficacy of the oral PanHER inhibitor PF-00299804 in patients with adenocarcinoma of the lung who are either non-smokers (<100 cigarette, cigar or pipe lifetime) or former light smokers ( less than 10 pack-years and stopped at least 15 years) or have known EGFR activating mutation; or patients with HER 2 amplification or mutation.

ELIGIBILITY:
Inclusion Criteria:

* Advanced adenocarcinoma of lung, measurable disease
* Non-smoker, or former light (less than 10 pack years and stopped at least 15 years); OR
* patients with known EGFR activating mutation regardless of smoking status
* ECOG(Eastern Cooperative Oncology Group) 0-1.

Cohort B (select sites only): patients with HER2 amplified or HER2 mutation-positive NSCLC; may have had prior therapy

Exclusion Criteria:

* Active brain metastases
* Prior systemic therapy for advanced disease in Cohort A only. Cohort B can have had any number of prior lines of systemic therapy.
* known EGFR wild type NSCLC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2009-03-11 (Actual); Primary Completion 2012-04-27 (Actual); Study Completion 2015-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (37):
- United States (28):
  - University of California, Irvine, Orange, California
  - Chao Family Comprehensive Cancer Center UC Irvine Medical Center, Orange, California
  - Bay Area Cancer Research Group, LLC, Pleasant Hill, California
  - Pacific Cancer Care, Salinas, California
  - San Francisco General Hospital, San Francisco, California
  - University of Colorado Clinical Trials Office (CTO), Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - Florida Cancer Specialists, Fort Myers, Florida
  - National Institutes of Health National Cancer Institute, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber Cancer lnstitute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - St. John's Hospital,, Springfield, Missouri
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Stony Brook University Medical Center - Cancer Center, Stony Brook, New York
  - Investigational Drug Service, Pharmacy Department, UNC Hospitals, Chapel Hill, North Carolina
  - Division of Hemotology/Oncology, Chapel Hill, North Carolina
  - UNC Hospitals, The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Morris Cancer Center, Durham, North Carolina
  - Legacy Pharma Research, Bismarck, North Dakota
  - Mid Dakota Clinic, P.C, Bismarck, North Dakota
  - Chattanooga Oncology & Hematology Associates, P.C., Chattanooga, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Virginia Cancer Institute, Richmond, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
- Hong Kong (3):
  - Department of Clinical Oncology, Tuen Mun Hospital, Tuenmen, NEW Territories
  - Department of Clinical Oncology, Tuen Mun Hospital, New Territories
  - Prince of Wales Hospital, Shatin, NT
- Japan (2):
  - The Cancer Institute Hospital of JFCR, Koto-Ku, Tokyo
  - Aichi cancer center central hospital Thoracic Oncology, Aichi
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University College of Medicine, Yonsei Cancer Center, Seoul
  - SamsungMedicalCenter, Sungkyunkwan Univ School of Medicine, Seoul
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Kris MG, Camidge DR, Giaccone G, Hida T, Li BT, O'Connell J, Taylor I, Zhang H, Arcila ME, Goldberg Z, Janne PA. Targeting HER2 aberrations as actionable drivers in lung cancers: phase II trial of the pan-HER tyrosine kinase inhibitor dacomitinib in patients with HER2-mutant or amplified tumors. Ann Oncol. 2015 Jul;26(7):1421-7. doi: 10.1093/annonc/mdv186. Epub 2015 Apr 21. PMID 25899785
- [Derived] Janne PA, Ou SI, Kim DW, Oxnard GR, Martins R, Kris MG, Dunphy F, Nishio M, O'Connell J, Paweletz C, Taylor I, Zhang H, Goldberg Z, Mok T. Dacomitinib as first-line treatment in patients with clinically or molecularly selected advanced non-small-cell lung cancer: a multicentre, open-label, phase 2 trial. Lancet Oncol. 2014 Dec;15(13):1433-1441. doi: 10.1016/S1470-2045(14)70461-9. Epub 2014 Nov 5. PMID 25456362
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A7471017&StudyName=Dacomitinib%20%28PF-00299804%29%20As%20A%20Single%20Oral%20Agent%20In%20Selected%20Patients%20With%20Adenocarcinoma%20Of%20The%20Lung%20%0A%20

RESULTS

PARTICIPANT FLOW:
Groups:
- Dacomitinib: Cohort A: Participants who had adenocarcinoma of lung, had not received prior systemic therapy and were either nonsmokers, former light smokers or were known to have an epidermal growth factor receptor (EGFR)-activating mutation, received dacomitinib 45 milligram (mg) or 30 mg tablet orally daily in cycles of 28 days until progression of disease, unacceptable toxicity, or participant withdrawal. Dose escalated to 45 mg in participants after at least 8 weeks of therapy who had started treatment at 30 mg and were tolerating treatment for at least 4 consecutive weeks as per investigator's judgment. Dose modifications for treatment-related toxicity were allowed for up to 2 dose reductions (to 30 mg and then to 15 mg) if the participant started at 45 mg. Dose interruption for treatment-related toxicity was also allowed as per investigator's discretion.
- Dacomitinib: Cohort B: Participants who had human epidermal growth factor receptor 2 (HER2) gene amplification or HER2 mutation, advanced non-small cell lung cancer (NSCLC) of any histology and had received prior chemotherapy or prior EGFR-targeted therapy, received dacomitinib 45 mg or 30 mg tablet orally daily in cycles of 28 days until progression of disease, unacceptable toxicity, or participant withdrawal. Participants who had not received prior therapy for advanced NSCLC, received 30 mg daily and participants who had received prior systemic therapy for advanced NSCLC, received 45 mg daily as starting dose. Dose escalated to 45 mg in participants after at least 8 weeks of therapy who had started treatment at 30 mg and were tolerating treatment for at least 4 consecutive weeks as per judgment of the investigator. Dose modifications for treatment-related toxicity were allowed for up to 2 dose reductions (to 30 mg and then to 15 mg) if the participant started at 45 mg.
Period: Overall Study
Arm/Group | Dacomitinib: Cohort A | Dacomitinib: Cohort B
Started | 89 | 30
Completed | 0 | 0
Not Completed | 89 | 30
Not completed — Death | 69 | 26
Not completed — Other | 5 | 0
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Adverse Event | 0 | 1
Not completed — Study terminated by sponsor | 11 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dacomitinib: Cohort A | Dacomitinib: Cohort B | Total
Number analyzed (Participants) | 89 | 30 | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (11.18) | 57.3 (10.88) | 61.3 (11.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 15 | 75
  Male | 29 | 15 | 44

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) at Month 4: Cohort A
Description: PFS at Month 4 was defined as percentage of participants who were alive and event free (event defined as progressive disease [PD] or death due to any cause, whichever occurs first) at 4 months after the first dose of study treatment. Documentation of progression was based on Response Evaluation Criteria in Solid Tumors version 1.0 (RECIST v1.0) criteria. PD = greater than or equal to (>=) 20 percent (%) increase in the sum of the longest dimensions of the target lesions taking as a reference the smallest sum of the longest dimensions recorded since the start of treatment, or the appearance of 1 or more new lesions, or unequivocal progression in non-target lesions.
Time Frame: Baseline up to Month 4
Population: As-enrolled population included all participants who were enrolled in the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dacomitinib: Cohort A
Number analyzed (Participants) | 89
percentage of participants | 76.9 [66.4 to 84.4]

2. Secondary Outcome: Progression-Free Survival (PFS) at Month 4: Cohort B
Description: PFS at Month 4 was defined as percentage of patients who were alive and event free (event defined as PD or death due to any cause, whichever occurs first) at 4 months after the first dose of study treatment. Documentation of progression was based on RECIST v1.0 criteria. PD: >=20% increase in the sum of the longest dimensions of the target lesions taking as a reference the smallest sum of the longest dimensions recorded since the start of treatment, or the appearance of 1 or more new lesions, or unequivocal progression in non-target lesions.
Time Frame: Baseline up to Month 4
Measure: Number (95% Confidence Interval); unit: percent chance of being event-free
Arm/Group | Dacomitinib: Cohort B
Number analyzed (Participants) | 30
percent chance of being event-free | 24.9 [11.0 to 41.7]

3. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time in months from the first dosing date to the date of first documentation of progression or death due to any cause, whichever occurs first. PFS was calculated as (first event date [if not reached, censored date as the last known event-free date] minus first dosing date plus 1) divided by 30.44. PD: >= 20% increase in the sum of the longest dimensions of the target lesions taking as a reference the smallest sum of the longest dimensions recorded since the start of treatment, or the appearance of 1 or more new lesions. Documentation of progression was determined from objective disease assessment based on RECIST v1.0 criteria.
Time Frame: Baseline until progression or initiation of new anti-cancer therapy or death, assessed at baseline, at the end of Cycle 1, Cycle 2, and then every other cycle.
Population: As-enrolled population included all participants who were enrolled in the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dacomitinib: Cohort A | Dacomitinib: Cohort B
Number analyzed (Participants) | 89 | 30
months | 11.5 [9.0 to 12.9] | 2.6 [1.8 to 3.7]

4. Secondary Outcome: Best Overall Response (BOR)
Description: BOR: best response recorded from treatment start until disease progression/recurrence based on RECIST v1.0. Complete Response (CR): disappearance of all lesions. Partial Response (PR): >=30% decrease in sum of longest diameters of target lesions taking as reference baseline sum of longest diameters, associated to non-progressive disease response for non target lesions. PD: >=20% increase in sum of longest diameters of target lesions taking as reference smallest sum of longest diameters since treatment start, or appearance of >=1 new lesion, or unequivocal progression in non-target lesions. Stable disease (SD): neither shrinkage for CR/PR nor increase for PD taking as reference smallest sum of longest diameters since treatment start. CR and PR had to be confirmed on a follow up imaging assessment >=4 weeks after the initial objective documentation of the response. SD must have met the SD criteria at least once after start of treatment in a minimum interval of 6 weeks.
Time Frame: as for outcome 3
Population: Response-evaluable population included all enrolled participants who received at least 1 dose of study medication, had an adequate baseline tumor assessment, and had at least 1 on-study tumor assessment after the first dosing.
Measure: Number; unit: participants
Arm/Group | Dacomitinib: Cohort A | Dacomitinib: Cohort B
Number analyzed (Participants) | 89 | 30
participants
  Complete Response | 1 | 0
  Partial Response | 47 | 3
  Stable Disease | 27 | 11
  Progressive Disease | 13 | 13
  Indeterminate | 1 | 3

5. Secondary Outcome: Duration of Response (DR)
Description: Time in months from the first documentation of objective tumor response to objective tumor progression or death due to any cause, whichever occurs first. Duration of tumor response was calculated as (the date of the first documentation of objective tumor progression or death due to any cause [if not reached, censored date] minus the date of the first CR or PR that was subsequently confirmed plus 1) divided by 30.44. DR was calculated for a subgroup of participants with a confirmed objective tumor response.
Time Frame: as for outcome 3
Population: DR was calculated for a subgroup of participants from the response-evaluable population, who had confirmed objective tumor response (CR or PR).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dacomitinib: Cohort A | Dacomitinib: Cohort B
Number analyzed (Participants) | 48 | 3
months | 12.9 [9.6 to 18.4] | 12.4 [11.0 to 13.9]

6. Secondary Outcome: Overall Survival (OS)
Description: Time in months from the start of study treatment to date of death due to any cause. OS was calculated as (the death date or last alive date minus the date of first dose of study medication plus 1) divided by 30.44. Death was determined from adverse event data (where outcome was death) or from follow-up contact data (where the participant current status was death).
Time Frame: Randomization until death or last date known to be alive.
Population: As-enrolled population included all participants who were enrolled in the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dacomitinib: Cohort A | Dacomitinib: Cohort B
Number analyzed (Participants) | 89 | 30
months | 29.5 [22.8 to 35.6] | 9.3 [6.6 to 20.8]

7. Secondary Outcome: European Organization for Research and Treatment of Cancer, Quality of Life Questionnaire Core-30 (EORTC QLQ-C30) Score
Description: EORTC QLQ-C30: included functional scales (physical, role, cognitive, emotional, and social), global health status (GHS), symptom scales (fatigue, pain, nausea/vomiting), and single items (dyspnea, appetite loss, insomnia, constipation, diarrhea, and financial difficulties). Most questions used 4- point scale (1 'Not at All' to 4 'Very Much'); 2 questions used 7-point scale (1 'Very Poor' to 7 'Excellent'). For GHS, functional scales, symptom scales and single items, scores were averaged, transformed to 0-100 scale; higher score=better level of functioning/health or greater degree of symptoms. Improvement was defined as a mean increase from baseline of ≥10 for GHS and functional scales or a mean decrease from baseline of ≤10 for symptom scales. Worsened was defined as a mean decrease from baseline of ≤10 for GHS and functional scales or a mean increase from baseline of ≥10 for symptom scales. Stable was a mean change from baseline of <10.
Time Frame: Baseline (Cycle [C]1 Day 1), up to C75
Population: Patient reported Outcome (PRO) analysis set:participants who received at least (>=) 1 dose of study medication (as-treated population), had baseline PRO assessments, >=1 on-study assessment submitted. 'N' (number of participants analyzed)=participants evaluable for this measure.n=participants evaluable at specified time points for given parameter.
Measure: Number; unit: number of participants
Arm/Group | Dacomitinib: Cohort A | Dacomitinib: Cohort B
Number analyzed (Participants) | 84 | 29
number of participants
  GHS: Improved | 22 | 3
  GHS: Worsened | 21 | 11
  GHS: Stable | 39 | 15
  Physical Functioning: Improved | 19 | 4
  Physical Functioning: Worsened | 22 | 7
  Physical Functioning: Stable | 42 | 18
  Role Functioning: Inproved | 24 | 7
  Role Functioning: Worsened | 30 | 10
  Role Functioning: Stable | 29 | 12
  Cognitive Functioning: Improved | 15 | 6
  Cognitive Functioning: Worsened | 24 | 9
  Cognitive Functioning: Stable | 44 | 14
  Emotional Functioning: Improved | 22 | 4
  Emotional Functioning: Worsened | 23 | 7
  Emotional Functioning: Stable | 38 | 18
  Social Functioning: Improved | 20 | 8
  Social Functioning: Worsened | 25 | 9
  Social Functioning: Stable | 37 | 12
  Fatigue: Improved | 30 | 7
  Fatigue: Worsened | 28 | 11
  Fatigue: Stable | 25 | 11
  Pain: Improved | 32 | 8
  Pain: Worsened | 24 | 11
  Pain: Stable | 27 | 10
  Nausea and Vomiting: Improved | 16 | 3
  Nausea and Vomiting: Worsened | 14 | 11
  Nausea and Vomiting: Stable | 53 | 15
  Dyspnea: Improved | 28 | 2
  Dyspnea: Worsened | 16 | 5
  Dyspnea: Stable | 39 | 22
  Appetite Loss: Improved | 22 | 3
  Appetite Loss: Worsened | 25 | 13
  Appetite Loss: Stable | 36 | 13
  Insomnia: Improved | 31 | 10
  Insomnia: Worsened | 19 | 5
  Insomnia: Stable | 33 | 14
  Constipation: Improved | 23 | 8
  Constipation: Worsened | 9 | 4
  Constipation: Stable | 50 | 17
  Diarrhea: Improved | 6 | 0
  Diarrhea: Worsened | 58 | 22
  Diarrhea: Stable | 19 | 7
  Financial Difficulties: Improved | 14 | 4
  Financial Difficulties: Worsened | 18 | 3
  Financial Difficulties: Stable | 51 | 22

8. Secondary Outcome: European Organization for Research and Treatment of Cancer, Quality of Life Questionnaire-Lung Cancer 13 (EORTC QLQ-LC13) Score
Description: QLQ-LC13 consisted of 13 questions relating to disease symptoms specific to lung cancer and treatment side effects typical of treatment with chemotherapy and radiotherapy experienced during past 1 week. The 13 questions comprised 1 multi-item scale for dyspnea and 10 single-item symptoms and side effects (coughing, hemoptysis, sore mouth, dysphagia, peripheral neuropathy, alopecia, chest pain, arm pain, other pain, and medicine for pain ). Response range: (1) not at all to (4) very much. Scores for each item were transformed to 0 to 100, where higher symptom score = greater degree of symptoms. Results are reported for coughing, hemoptysis, sore mouth, dysphagia, peripheral neuropathy, alopecia, chest pain, arm pain, and other pain. Improvement was defined as a mean decrease from baseline of ≤10. Worsened was defined as a mean increase from baseline of ≥10. Stable was a mean change from baseline of <10.
Time Frame: Baseline (C1D1) up to C75
Population: PRO analysis set: participants who received >=1 dose of study medication (as-treated population), had baseline PRO assessments, >=1 on-study assessment submitted. n=participants evaluable at specified time points for given parameter.
Measure: Number; unit: number of participants
Arm/Group | Dacomitinib: Cohort A | Dacomitinib: Cohort B
Number analyzed (Participants) | 84 | 29
number of participants
  Dyspnoea: Improved | 21 | 5
  Dyspnoea: Worsened | 16 | 8
  Dyspnoea: Stable | 47 | 16
  Coughing: Improved | 36 | 12
  Coughing: Worsened | 11 | 4
  Coughing: Stable | 37 | 13
  Haemoptysis: Improved | 4 | 1
  Haemoptysis: Worsened | 2 | 2
  Haemoptysis: Stable | 78 | 26
  Sore Mouth: Improved | 5 | 2
  Sore Mouth: Worsened | 45 | 18
  Sore Mouth: Stable | 34 | 9
  Dysphagia: Imporved | 8 | 2
  Dysphagia: Worsened | 13 | 7
  Dysphagia: Stable | 63 | 19
  Peripheral Neuropathy: Improved | 11 | 6
  Peripheral Neuropathy: Worsened | 28 | 8
  Peripheral Neuropathy: Stable | 45 | 15
  Alopecia: Improved | 6 | 10
  Alopecia: Worsened | 35 | 2
  Alopecia: Stable | 42 | 16
  Pain in Chest: Improved | 26 | 7
  Pain in Chest: Worsened | 11 | 5
  Pain in Chest: Stable | 47 | 16
  Pain in Arm or Shoulder: Improved | 23 | 5
  Pain in Arm or Shoulder: Worsened | 14 | 5
  Pain in Arm or Shoulder: Stable | 47 | 18
  Pain in Other Parts: Improved | 28 | 7
  Pain in Other Parts: Worsened | 20 | 9
  Pain in Other Parts: Stable | 33 | 12

9. Secondary Outcome: Trough Plasma Concentrations (Ctrough) of Dacomitinib
Description: Results for Ctrough were summarized as per the dose received during given cycle: no dose (treatment interruption at any cycle due to treatment-related toxicity), dacomitinib 15 mg (dacomitinib 15 mg at any cycle due to treatment-related toxicity at higher doses), 30 mg (dacomitinib 30 mg at any cycle as starting dose or dose reduction due to treatment-related toxicity at higher doses), 45 mg (dacomitinib 45 mg at any cycle as starting dose or dose escalation due to satisfactory toleration of dacomitinib 30 mg treatment).
Time Frame: Predose on C1D14, C2D1, C3D1, C4D1
Population: Pharmacokinetic (PK) analysis set: all participants who received at least 1 dose of study medication at selected PK sites from whom at least 1 PK sample were obtained. 'N' (number of participants analyzed) = participants who were evaluable for this measure at any time point. n = participants evaluable at given time points for specified dose.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Dacomitinib: Cohort A | Dacomitinib: Cohort B
Number analyzed (Participants) | 84 | 30
nanogram per milliliter (ng/mL)
  C1D14: No Dose (Cohort A n=5; Cohort B n=5) | 48.30 (53.225) | 52.04 (26.656)
  C1D14: 30 mg (Cohort A n=28; Cohort B n=2) | 56.61 (25.795) | NA (NA) — Mean and standard deviation of fewer than 3 participants was not considered meaningful, hence not summarized.
  C1D14: 45 mg (Cohort A n=51; Cohort B n=20) | 76.50 (30.261) | 74.22 (27.617)
  C2D1: No Dose (Cohort A n=4; Cohort B n=2) | 27.41 (19.526) | NA (NA) — Mean and standard deviation of fewer than 3 participants was not considered meaningful, hence not summarized.
  C2D1: 15 mg (Cohort A n=1; Cohort B n=0) | NA (NA) — Mean and standard deviation of fewer than 3 participants was not considered meaningful, hence not summarized. | NA (NA) — Mean and standard deviation of fewer than 3 participants was not considered meaningful, hence not summarized.
  C2D1: 30 mg (Cohort A n=31; Cohort B n=6) | 54.45 (22.120) | 51.78 (21.027)
  C2D1: 45 mg (Cohort A n=42; Cohort B n=11) | 69.98 (26.899) | 79.63 (22.437)
  C3D1: No Dose (Cohort A n=5; Cohort B n=1) | 41.80 (32.179) | NA (NA) — Mean and standard deviation of fewer than 3 participants was not considered meaningful, hence not summarized.
  C3D1: 15 mg (Cohort A n=2; Cohort B n=0) | NA (NA) — Mean and standard deviation of fewer than 3 participants was not considered meaningful, hence not summarized. | NA (NA) — Mean and standard deviation of fewer than 3 participants was not considered meaningful, hence not summarized.
  C3D1: 30 mg (Cohort A n=31; Cohort B n=4) | 49.13 (19.726) | 58.43 (21.009)
  C3D1: 45 mg (Cohort A n=31; Cohort B n=8) | 73.03 (35.452) | 84.67 (34.287)
  C4D1: No Dose (Cohort A n=3; Cohort B n=1) | 37.80 (24.908) | NA (NA) — Mean and standard deviation of fewer than 3 participants was not considered meaningful, hence not summarized.
  C4D1: 15 mg (Cohort A n=6; Cohort B n=0) | 21.92 (6.7514) | NA (NA) — Mean and standard deviation of fewer than 3 participants was not considered meaningful, hence not summarized.
  C4D1: 30 mg (Cohort A n=33; Cohort B n=2) | 55.27 (20.856) | NA (NA) — Mean and standard deviation of fewer than 3 participants was not considered meaningful, hence not summarized.
  C4D1: 45 mg (Cohort A n=25; Cohort B n=7) | 56.02 (23.749) | 83.57 (48.302)
  C2D1: 25 mg (Cohort A n=0; Cohort B n=1) | NA (NA) — Mean and standard deviation of fewer than 3 participants was not considered meaningful, hence not summarized. | NA (NA) — Mean and standard deviation of fewer than 3 participants was not considered meaningful, hence not summarized.

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Dacomitinib: Cohort A | Dacomitinib: Cohort B
Serious Adverse Events (participants affected / at risk) | 29/89 | 9/30
Other Adverse Events (participants affected / at risk) | 89/89 | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dacomitinib: Cohort A (N=89) | Dacomitinib: Cohort B (N=30)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Haemorrhagic arteriovenous malformation (Congenital, familial and genetic disorders) | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 3
Dysphagia (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 2
Stomatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2
Asthenia (General disorders) | 3 | 0
Disease progression (General disorders) | 2 | 1
Pyrexia (General disorders) | 1 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 1
Infection (Infections and infestations) | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Paronychia (Infections and infestations) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Colon cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 1
Confusional state (Psychiatric disorders) | 2 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Vasculitis (Vascular disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Transaminases (Investigations) | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dacomitinib: Cohort A (N=89) | Dacomitinib: Cohort B (N=30)
Anaemia (Blood and lymphatic system disorders) | 5 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 2 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 2 | 0
External ear pain (Ear and labyrinth disorders) | 1 | 0
Hearing impaired (Ear and labyrinth disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Blepharitis (Eye disorders) | 1 | 0
Chalazion (Eye disorders) | 1 | 0
Conjunctivitis (Infections and infestations) | 4 | 0
Dry eye (Eye disorders) | 18 | 2
Eye irritation (Eye disorders) | 3 | 1
Eye oedema (Eye disorders) | 2 | 0
Eye pain (Eye disorders) | 3 | 0
Eye pruritus (Eye disorders) | 3 | 1
Eye swelling (Eye disorders) | 1 | 0
Eyelash thickening (Eye disorders) | 1 | 0
Eyelid pain (Eye disorders) | 1 | 0
Growth of eyelashes (Eye disorders) | 2 | 0
Keratitis (Eye disorders) | 1 | 0
Lacrimation increased (Eye disorders) | 6 | 0
Ocular hyperaemia (Eye disorders) | 1 | 1
Trichiasis (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 6 | 2
Visual impairment (Eye disorders) | 2 | 0
Vitreous floaters (Eye disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 6 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 8 | 2
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 3 | 0
Anorectal disorder (Gastrointestinal disorders) | 1 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 2 | 0
Cheilitis (Gastrointestinal disorders) | 8 | 4
Constipation (Gastrointestinal disorders) | 13 | 9
Defaecation urgency (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 85 | 28
Dry mouth (Gastrointestinal disorders) | 14 | 4
Duodenitis (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 4 | 2
Dysphagia (Gastrointestinal disorders) | 2 | 1
Faecal incontinence (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 2 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 3
Gingival bleeding (Gastrointestinal disorders) | 4 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0
Gingivitis (Infections and infestations) | 1 | 0
Glossitis (Gastrointestinal disorders) | 1 | 0
Glossodynia (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 2 | 0
Haematochezia (Gastrointestinal disorders) | 2 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 3 | 1
Haemorrhoids (Gastrointestinal disorders) | 8 | 1
Lip disorder (Gastrointestinal disorders) | 1 | 0
Lip pain (Gastrointestinal disorders) | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 25 | 12
Oral discomfort (Gastrointestinal disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0
Paraesthesia oral (Gastrointestinal disorders) | 1 | 0
Periodontal disease (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 35 | 6
Swollen tongue (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 20 | 9
Adverse drug reaction (General disorders) | 1 | 0
Asthenia (General disorders) | 3 | 1
Axillary pain (General disorders) | 1 | 0
Catheter site related reaction (General disorders) | 1 | 0
Chest discomfort (General disorders) | 4 | 1
Chest pain (General disorders) | 9 | 1
Chills (General disorders) | 3 | 1
Face oedema (General disorders) | 1 | 1
Fatigue (General disorders) | 36 | 17
Gait disturbance (General disorders) | 1 | 0
Influenza like illness (General disorders) | 1 | 0
Infusion site extravasation (General disorders) | 1 | 0
Local swelling (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Mucosal dryness (General disorders) | 1 | 1
Mucosal inflammation (General disorders) | 28 | 11
Nodule (General disorders) | 1 | 0
Oedema (General disorders) | 2 | 1
Oedema peripheral (General disorders) | 9 | 2
Pain (General disorders) | 6 | 0
Pyrexia (General disorders) | 4 | 1
Xerosis (General disorders) | 7 | 4
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Seasonal allergy (Immune system disorders) | 1 | 0
Abscess limb (Infections and infestations) | 1 | 0
Bacterial disease carrier (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 3 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 1
Cystitis (Infections and infestations) | 1 | 0
Ear infection (Infections and infestations) | 1 | 0
Eye infection (Infections and infestations) | 1 | 1
Folliculitis (Infections and infestations) | 6 | 0
Fungal infection (Infections and infestations) | 4 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Laryngitis (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 2 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Myringitis (Infections and infestations) | 1 | 0
Nasal vestibulitis (Infections and infestations) | 2 | 2
Nasopharyngitis (Infections and infestations) | 6 | 0
Oral herpes (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 1 | 0
Paronychia (Infections and infestations) | 35 | 10
Pharyngitis (Infections and infestations) | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Pyoderma (Infections and infestations) | 1 | 0
Rash pustular (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0
Skin candida (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 2 | 3
Staphylococcal infection (Infections and infestations) | 1 | 0
Tinea pedis (Infections and infestations) | 3 | 0
Upper respiratory tract infection (Infections and infestations) | 9 | 2
Urinary tract infection (Infections and infestations) | 8 | 2
Viral infection (Infections and infestations) | 2 | 0
Viral upper respiratory tract infection (Infections and infestations) | 3 | 0
Vulvitis (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 3 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Osteoradionecrosis (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Scratch (Injury, poisoning and procedural complications) | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 3 | 3
Aspartate aminotransferase increased (Investigations) | 3 | 3
Blood alkaline phosphatase increased (Investigations) | 2 | 5
Blood creatine phosphokinase (Investigations) | 1 | 0
Blood uric acid increased (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Protein total decreased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 8 | 4
Weight increased (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 28 | 9
Dehydration (Metabolism and nutrition disorders) | 8 | 6
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 14 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 4 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 15 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 9 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 3
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dizziness (Nervous system disorders) | 7 | 0
Dysgeusia (Nervous system disorders) | 14 | 6
Headache (Nervous system disorders) | 15 | 2
Hypoaesthesia (Nervous system disorders) | 3 | 0
Memory impairment (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 2 | 2
Paraesthesia (Nervous system disorders) | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 8 | 3
Restless legs syndrome (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Tension headache (Nervous system disorders) | 2 | 0
Tremor (Nervous system disorders) | 2 | 1
Anxiety (Psychiatric disorders) | 3 | 0
Depressed mood (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 2 | 1
Insomnia (Psychiatric disorders) | 10 | 2
Mood swings (Psychiatric disorders) | 1 | 0
Bladder discomfort (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 4 | 1
Haematuria (Renal and urinary disorders) | 2 | 2
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0
Polyuria (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Pyuria (Infections and infestations) | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 2 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0
Menstruation irregular (Reproductive system and breast disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 2 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 28 | 11
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 | 5
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 21 | 5
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 10 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 11 | 2
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 13 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acne (Skin and subcutaneous tissue disorders) | 18 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 12 | 5
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 2 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 3 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 68 | 22
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 39 | 15
Eczema (Skin and subcutaneous tissue disorders) | 2 | 0
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 6 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 7 | 1
Exfoliative rash (Skin and subcutaneous tissue disorders) | 10 | 0
Hair colour changes (Skin and subcutaneous tissue disorders) | 1 | 0
Hair disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 5 | 0
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 1 | 0
Hirsutism (Skin and subcutaneous tissue disorders) | 4 | 0
Hypertrichosis (Skin and subcutaneous tissue disorders) | 2 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 1 | 1
Nail bed bleeding (Skin and subcutaneous tissue disorders) | 1 | 0
Nail bed inflammation (Skin and subcutaneous tissue disorders) | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 19 | 2
Nail dystrophy (Skin and subcutaneous tissue disorders) | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 2 | 0
Onycholysis (Skin and subcutaneous tissue disorders) | 3 | 0
Onychomadesis (Skin and subcutaneous tissue disorders) | 2 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 2
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 19 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 0
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 22 | 12
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 6 | 3
Rash erythematous (Skin and subcutaneous tissue disorders) | 5 | 5
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1
Scab (Skin and subcutaneous tissue disorders) | 1 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 3 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2 | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 20 | 7
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 3 | 1
Skin mass (Skin and subcutaneous tissue disorders) | 2 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Telangiectasia (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 4 | 0
Embolism (Vascular disorders) | 1 | 0
Flushing (Vascular disorders) | 3 | 0
Haematoma (Vascular disorders) | 1 | 0
Hot flush (Vascular disorders) | 2 | 0
Hypertension (Vascular disorders) | 6 | 0
Hypotension (Vascular disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Eyelids pruritus (Eye disorders) | 0 | 1
Glaucoma (Eye disorders) | 0 | 1
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1
Chapped lips (Gastrointestinal disorders) | 0 | 1
Lip dry (Gastrointestinal disorders) | 0 | 2
Oral mucosal erythema (Gastrointestinal disorders) | 0 | 1
Early satiety (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Ulcer (General disorders) | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 1
Blood bilirubin (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 1
International normalised ratio increased (Investigations) | 0 | 1
Prothrombin time prolonged (Investigations) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Soft tissue disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 1
Drooling (Nervous system disorders) | 0 | 1
Mood altered (Psychiatric disorders) | 0 | 1
Nocturia (Renal and urinary disorders) | 0 | 1
Dyspareunia (Reproductive system and breast disorders) | 0 | 1
Vaginal discharge (Reproductive system and breast disorders) | 0 | 1
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1
Deafness unilateral (Ear and labyrinth disorders) | 1 | 0
Conjunctival hyperaemia (Eye disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 1
Peripheral swelling (General disorders) | 2 | 2
Diverticulitis (Infections and infestations) | 1 | 0
Nail infection (Infections and infestations) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 1
Blood creatinine increased (Investigations) | 0 | 1
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Irritability (Psychiatric disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal ulceration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Results have been included for Cohort B and updated for Cohort A since the Primary completion date.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.